CLINICAL TRIAL: NCT00936026
Title: Open, Single Center, Three Periods, Fixed Sequence Design Study on the Effects of Clopidogrel Co-administration on the Pharmacokinetics of Neramexane
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Dr. med. Margarete Müller, AAIPharma Deutschland gmbH & Co. KG
Masking: None
Other Study IDs: MRZ 92579/TI/1002
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2009-07

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — neramexane

INTERVENTIONS:
Drug: Neramexane — Drug-Drug Interaction Study

SUMMARY:
Primary:

To assess the effects of CYP2B6 inhibition by repeated dose Clopidogrel (75 mg/day) co-administration on the single-dose pharmacokinetics of Neramexane

Secondary:

To assess safety and tolerability of Neramexane single dose treatment alone and co-administration of a Neramexane single-dose with a Clopidogrel repeated dose treatment

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult subject of white origin, who is able to read, to write and fully understand German language
2. Aged 18 to 45 years
3. BMI of 18-28 kg/m2 and a body weight of 50-90 kg
4. Willing and able to provide written informed consent after having been informed of the requirements and the restrictions of the study. Female subjects of childbearing potential must agree to use a highly effective method of birth control defined as those which result in a low failure rate (i.e. less than 1 % per year) when used consistently and correctly such as sexual abstinence, vasectomised partner, non hormonal IUDs, double barrier methods, for instance, e.g. condom and spermicide cream.

Exclusion Criteria:

1. History of clinically relevant allergy or known hypersensitivity to Neramexane/ Memantine/Amantadine and their derivatives
2. History of clinically relevant allergy or known hypersensitivity to Clopidogrel
3. Exposure to another investigational agent within the last two months before Day 1 of Period 1
4. History of clinically relevant allergy or known hypersensitivity to any inactive ingredient in any of the used investigational products or the metabolic inhibitor
5. Lactating or pregnant females or females planning to become pregnant during study conduct or within 2 months after end of study
6. Any contraindications which are indicated in the topically valid SPC for Plavix®: severe hepatic impairment; active pathological bleeding such as peptic ulcer or intracranial hemorrhage

   Lack of suitability for the trial:
7. Any evidence of a significant cardiovascular, pulmonary, renal, hepatic, gastrointestinal, endocrinological, metabolic or other disease at screening
8. History of malignancy
9. Any clinically relevant deviation in clinical or laboratory assessment
10. ECG abnormalities of clinical relevance, in particular abnormal prolongations of QT/QTc-interval (i.e. QTc ≥ 450 ms, PQ ≥ 220 ms)
11. Systolic blood pressure <95 mmHg or >150 mmHg or diastolic blood pressure < 50 mmHg or >90 mmHg in supine position
12. Pulse rate <45 or >100 beats per minute
13. Chronic or acute clinically relevant infections
14. Acute or chronic disease, especially psychiatric or neurologic disorders
15. History of alcohol or drug dependence
16. Alcohol consumption averaging more than 40 g for male and more than 20 g for female subjects daily within the last year
17. Regular caffeine consumption averaging more than 1 L of coffee and/or tea daily or more than 1 L of caffeine-containing lemonades per day within the last year
18. Disorders or surgery of the gastrointestinal tract which may interfere with drug absorption or may otherwise influence the pharmacokinetics of the investigational medicinal products (e.g. cholecystectomy, ulcus, etc.)
19. Anticipated donation of spermatocytes or oocytes for medically assisted reproduction techniques [ART] within two months after the last dose of the present study
20. Use of any prescribed medication for four weeks prior to the first administration of IMP.

    * Regular use of over-the-counter drugs in the 4 weeks prior to the first administration of the IMP
    * Occasional use of OTC drugs (except paracetamol, maximum 1 g/day) within the 2 weeks prior to the first administration of the IMP.
    * Stable intake of thyroid hormone substitution will be allowed.
21. Use of any food, food supplement or medication known to induce or inhibit CYP3A4 or other cytochrome P450 enzymes within two weeks preceding the start of the study (Day 1), e.g. grapefruit, St. John's wort
22. Female subjects who employed any form of hormonal contraception within 2 months prior to study Day 1 (e.g. oral contraceptives, hormone releasing intrauterine contraceptive devices [IUDs], etc.)
23. Consumption of xanthine derivates (including caffeine) within two days prior to Day 1
24. Smoker and user of snuff, nicotine replacement and chewing tobacco
25. Previous enrolment into the clinical phase of the current study
26. Positive results in any of the serology tests
27. Blood donation more than 450 mL within 60 days prior to Day 1
28. Positive pregnancy test, if female
29. Positive drug screen or alcohol test

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- AAIPharma Deutschland gmbH & Co. KG, Neu-Ulm, Bavaria, Germany